CLINICAL TRIAL: NCT05261022
Title: Love Together, Parent Together (L2P2): A Protocol for a Pilot RCT of a Brief Writing Intervention for Interparental Couples With Young Children Amid the COVID-19 Pandemic
Brief Title: Love Together, Parent Together: A Protocol for a Pilot Study of an Intervention for Interparental Couples With Young Children
Acronym: L2P2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: York University (Other)
Collaborators: University of Toronto (Other); McMaster University (Other)
Responsible Party: Principal Investigator, Heather Prime, Assistant Professor, York University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: e2022-267
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Interparental Conflict; Marital Conflict; Marital Relationship; Internet-Based Intervention; Family Conflict
Keywords: Online Intervention; Family Systems; Randomized Controlled Trial; Writing Intervention; Couples' relationships

STUDY DESIGN:
Intervention Model Description: The current study is a two-arm (intervention vs. waitlist) design with pre-, 1-week post-, and 1- and 3-month follow-up assessments. The first 120 interparental couples who meet eligibility criteria and consent will be included in the study. The entirety of the study will be conducted online (via mobile or computer). The writing assignments (intervention vs. inactive-control task) will commence approximately one week following baseline surveys, which will include three writing sessions over the course of 12 weeks (one session every 4 weeks). Following the 3 month follow-up, couples randomised to the waitlist control condition will be invited to participate in the writing program (i.e., three writing sessions over the course of 12 weeks).
Who Masked: Investigator
Masking Description: Participants will be unmasked to their group assignment as they will be told their group assignment, by virtue of the psychosocial intervention. There is no care provider (the intervention is participant-directed and fully online). Participants report on their own outcomes and thus outcomes are not masked. Feasibility outcomes are masked. Study team investigators, including data analysts, will be masked. The research coordinator will be the only unmasked member of the research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Love Together, Parent Together Intervention (Experimental): Participants will take part in a 3-session writing intervention over the course of 12-week. They will complete a fact-based summary of a recent conflict and answer questions on conflict/conflict-related distress. Next, they will be asked to complete a 9-minute writing task where they reappraise the conflict they previously reported. First, they will watch an instructional video of how to engage in the writing task, by providing definitions and examples of potentially useful conflict reappraisal strategies. Writing prompts include: "… Think about this disagreement … from the perspective of a neutral third party who wants the best for all involved…"; "…what obstacles do you face in trying to take this perspective…?";"… How might you be most successful in taking this perspective … over the next 2 weeks?" Participants in the intervention group will receive emails to prompt use of the reappraisal strategy between writing sessions.
  Interventions: Behavioral: Love Together, Parent Together (L2P2)
- Wait-List Control Group (No Intervention): Participants will take part in a waitlist control group. They will participate in the same number of assessment/sessions as the experimental group. In the sessions that correspond to the intervention (one session every 4 weeks over the course of 12 weeks as in the intervention group), the waitlist group will complete a basic writing task (identical to the intervention group, wherein they provide a fact-based summary of a recent conflict) and they will complete questions regarding conflict history and conflict-related distress. No other writing tasks will take place.
  Following the 3-month assessment, they will be offered the writing intervention.

INTERVENTIONS:
Behavioral: Love Together, Parent Together (L2P2) — Love Together Parent Together (L2P2) is a brief, low-intensity relationship intervention intended to improve the interparental relationship for parents of young children.
  Other Names: L2P2
  Arms: Love Together, Parent Together Intervention

SUMMARY:
The COVID-19 pandemic has created a population-level threat to social relationships that requires a population-level solution. Among those who are particularly vulnerable to heightened conflict are interparental couples with young children, whose relationships may have already been under pressure prior to the pandemic. Reduced couples' satisfaction has been reported since the start of the pandemic, with over one-third of romantic partners reporting heightened conflict due to COVID-19. Couples are likely to stay in disharmonious relationships during times of socioeconomic upheaval, with the potential for relationship problems to persist over time. This may have serious implications for the mental health of parents, parent-child relationships, and children's emotional and behavioural problems (EBPs). Such a pattern is a societal concern given the known associations between couples' relationship quality and a number of critical indicators of population health, such as intimate partner violence, physical health and all-cause mortality, and economic instability, particularly for women. The current study protocol is for a pilot randomized controlled trial (RCT) of the Love Together Parent Together (L2P2) program-a brief, low-intensity, scalable relationship intervention for parents of young children. The two-arm (treatment vs. waitlist) pilot RCT will assess the feasibility goals: continued relationship-building with established recruitment partners and outreach to additional recruitment partners to increase enrolment rates; recruitment of a diverse sample in terms of sociocultural identity factors, pandemic-related stress, and relationship distress; acceptability of randomization; outcome assessment schedule completion (for treatment and control groups), retention and adherence to the program; and program acceptability. Additionally, the investigators will conduct a preliminary evaluation of treatment effects by examining group differences in couples-focused (i.e., couples' relationship, conflict-related negativity, interparental functioning) and family-focused outcomes (i.e., parent-child relations, parent mental health and child outcomes). A scalable couples-focused intervention is critically needed to circumvent the social consequences of the pandemic on young families.

ELIGIBILITY:
Inclusion Criteria:

* Both participants endorse being in a relationship
* Both partners reside in the same house
* There are one or more children under the age of 6 living at home
* Both participants are over age 18 years
* Both members of a couple agree to participate

Exclusion Criteria:

- No current plans or history of separation or divorce

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Risk for Relationship Distress - Dyadic Adjustment Scale | Week 0-22
  The percentage of participants scoring in the 'clinical range' (<13) on the Dyadic Adjustment Scale. Minimum score=1, maximum score=22. Lower scores correspond to worse outcomes.
Risk for Relationship Distress - COVID-19 Family Stressors | Week 0
  The percentage of participants scoring 'high' (>29) on the COVID-19 Family Stressor Scale. Minimum score=16, maximum score=48. Higher scores correspond to worse outcomes.
COVID Coping/Benefits | Week 0
  Background information. Minimum score=14, maximum score=42 . Higher scores correspond to better outcomes.
Adverse Childhood Experiences | Week 0
  Background information. Adverse Childhood Experiences Scale. Minimum score=0, maximum score=14. Higher scores correspond to higher ACES count.
Participants Enrolled Per Week | Week 0
  Number of participants enrolled per week, stratified by recruitment source.
Participant Education | Week 0
  The percentage of participants with less than or equal to a College degree.
Participant Income | Week 0
  The percentage of participants income that is less than or equal to the regional median.
Racial Diversity | Week 0
  The percentage of participants who identify as part of a racialized group.
Sexual Diversity | Week 0
  The percentage of participants who are gender and/or sexually diverse.
Immigration Status | Week 0
  The percentage of participants who were born outside of Canada.
Adherence | Week 1-9
  The percentage of participants who complete 2/3 intervention sessions.
Acceptability | Week 10
  The percentage of participants reporting at least 'agree' on scales of attitude, burden, perceived effectiveness, and ethicality on the Implementation Acceptability Scale. Minimum score=7, maximum score=35. Higher scores correspond to higher acceptability.
Uptake | Week 5-22
  The percentage of participants reporting some use of conflict reappraisal outside of intervention sessions (i.e., reporting a score of 3 or more on a scale of 1-7). Minimum score=1, maximum score=7. Higher scores correspond to better outcomes.
Retention | Week 22
  The percentage of participants who complete their Randomly Allocated Assignment (defined as completing baseline, 2/3 writing sessions, post-intervention, and 1/2 follow-up surveys).

SECONDARY OUTCOMES:
Couples' Relationship Quality | Week 0-22
  Using the Perceived Relationship Quality Scale. Minimum score=18, maximum score=126. Higher scores correspond to better outcomes.
Conflict Frequency | Week 0-22
  Using one item on a 7-point Likert scale: "Think about your experiences with your partner over the last four weeks. How often did you and your partner argue with each other?" Minimum score=1, maximum score=7. Higher scores correspond to worse outcomes.
Conflict-Related Negativity | Week 1-9
  Using two items following a fact-based summary: "I was angry at my partner for his/her behaviour during this conflict," "My partner's behaviour during this conflict was highly upsetting to me." Minimum score=2, maximum score=14. Higher scores correspond to worse outcomes.
Coparenting | Week 0-22
  The Brief Coparenting Relationship Scale. Minimum score=0, maximum score=84. Higher scores correspond to better outcomes.
Brief Coparenting Assessment | Week 1-9
  Six items from the Brief Coparenting Relationship Scale (Feinberg et al., 2012). Minimum score = 0, maximum score = 36. Higher scores correspond to better outcomes.
Parent-Child Positivity | Week 0-22
  Using the 5-item parent-reported positivity subscale of the Parenting Practices Scale. Minimum score=5, maximum score=25. Higher scores correspond to better outcomes.
Parent-Child Negativity | Week 0-22
  Using the 5-item parent-reported negativity subscale of the Parenting Practices Scale. Minimum score=5, maximum score=25. Higher scores correspond to worse outcomes.
Parent Mental Health | Week 0-22
  Using the Kessler Psychological Distress Scale. Minimum score=10, maximum score=50. Higher scores correspond to worse outcomes.
Perceived Partner Responsiveness | Week 0-22
  Using the Perceived Partner Responsiveness-Insensitivity Scale (PRI-R)- Brief Version. Minimum score=8, maximum score=40. Higher scores correspond to better outcomes.
Responsiveness Towards Partner | Week 0-22
  Using the Perceived Partner Responsiveness-Insensitivity Scale (PRI) - Brief with items flipped to reflect responsiveness towards partner. Minimum score=8, maximum score=40. Higher scores correspond to better outcomes.
Family Functioning | Week 0-22
  Using the Family Assessment Device. Minimum score=12, maximum score=48. Higher scores correspond to worse outcomes.
Child Emotional and Behavioural Problems | Week 0-22
  Scores will be standardized within each age group and used as a single outcome variable.
  Using the Pediatric Symptom Checklist (Baby, Preschool and Standard versions). The Baby Pediatric Symptom Checklist: minimum score=0, maximum score=26. Higher scores correspond to worse outcomes.
  The Preschool Pediatric Symptoms Checklist (PPSC-17): minimum score=0, maximum score=36. Higher scores correspond to worse outcomes.
  The Pediatric Symptom Checklist-17: minimum score=0, maximum score=34. Higher scores correspond to worse outcomes.
Child Effortful Control | Week 0-22
  Using the Effortful Control subscale (12 items) of the Infant Behaviour Questionnaire- Revised Very Short Form (3-12 months), Early Childhood Behavior Questionnaire-Revised Very Short Form (18-36 months) and Children's Behaviour Questionnaire-Revised Very Short Form (3-7 years). Minimum score=0 , maximum score=84. Higher scores correspond to better outcomes.
Child Development | Week 0-22
  Using the 10-item Developmental Milestones scale from The Survey of Well-being of Young Children (i.e., the 2, 4, 6, 9, 12, 15, 18, 24, 30, 36, 48 and 60 month age-specific forms). Minimum score=0, maximum score =20. Higher scores correspond to better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Prime, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided